CLINICAL TRIAL: NCT01608893
Title: Carvedilol for Prevention of Paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Libin Cardiovascular Institute of Alberta (Other)
Responsible Party: Principal Investigator, Dr. Anne M. Gillis, Professor of Medicine, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Carvedilol for PAF
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoprolol (Active Comparator): The metoprolol arm patients are stratified by the arrhythmia management strategy Rate or Rhythm control and metoprolol is dose titrated from 25 mg bid to a maximum of 50 mg bid over one month then patients are followed for 6 months.
  Interventions: Drug: Metoprolol
- Carvedilol (Active Comparator): The carvedilol arm patients are stratified by the arrhythmia management strategy Rate or Rhythm control and carvedilol is dose titrated from 3.25 mg bid to maximum dose of 25 mg bid over one month then patients are followed for 6 months.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — 6.25 po bid titrated to 25 mg bid as tolerated over a 1 month period
  Other Names: Coreg
  Arms: Carvedilol
Drug: Metoprolol — titrated to 50 mg po bid as tolerated over a 1 month period
  Other Names: Lopressor
  Arms: Metoprolol

SUMMARY:
Atrial fibrillation (AF) is the most common sustained heart rhythm disorder and is associated with significant symptoms and health problems including an increased risk of stroke and death. Current drug therapies are often ineffective and associated with significant side effects. Abnormalities of calcium regulation in cells may lead to triggers for AF. Emerging data suggest that abnormal intracellular calcium regulation mediated through the ryanodine receptor in heart cells may contribute to AF. Recently the investigators have shown that the β-blocker carvedilol which is most commonly used to treat patients with heart failure, modifies calcium regulation mediated through the ryanodine receptor. At present this drug is not frequently used to treat AF. Therefore the investigators will conduct a randomized trial comparing carvedilol to metoprolol for prevention of paroxysmal AF. This may result in improved health and quality of life for people who suffer AF.

DETAILED DESCRIPTION:
The study population will consist of patients with electrocardiographically documented symptomatic paroxysmal AF (≥ 2 episodes of ≥ 15 min duration within a six month period) while on stable antiarrhythmic drug therapy. Patients will be excluded if they have AF due to a reversible cause, persistent AF, significant heart failure or a life expectancy of less than one year. Eligible patients will be randomized to carvedilol or metoprolol and followed for 13 months. Randomization will be stratified based on the AF management strategy (rate or rhythm control). Carvedilol and metoprolol will be initiated over a one month drug titration period to achieve doses of 25mg bid and 50 mg bid respectively. AF occurrence will be documented using event recorders. The co-primary outcome measures are survival free from AF after one month blanking period for drug titration and the number of days in AF detected during follow-up. Secondary outcomes include event free survival to first symptomatic episode of AF, days in symptomatic AF, time between first and second episodes of AF, proportion of patients who develop persistent AF, AF Severity Scale, CCS-AF symptom score, ventricular rate during AF, proportion of patients with discontinuation of the assigned therapy and number of emergency department visits or hospitalizations for cardiovascular causes. Adverse effects and need to discontinue carvedilol or metoprolol will be documented. This study will determine whether carvedilol is safe and effective for prevention of recurrent paroxysmal AF in a general population with AF. Data will be analyzed on an intention to treat basis. Three hundred patients will be recruited over 4 years. The sample size is based on an estimated 20% reduction in event free survival from AF (power 0.90, α = 0.05). Patients will be recruited from our AF clinic population which averages 50 new referrals per month and over 2500 referrals since it's' inception in 2005.

ELIGIBILITY:
Inclusion Criteria:

* Must be in sinus rhythm at enrollment
* ECG documented symptomatic PAF (> 2 episodes of > 15minutes duration over a 6 month period)

Exclusion Criteria:

* AF due to reversible causes
* Contraindication or previous significant adverse reaction to Beta blocker therapy
* Persistent AF
* NYHA Class II or greater CHF
* LVEF < or = 35%
* Life expectancy < 1 year
* Geographic isolation
* Unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival to first detected AF after the one month blanking period for dose titration | 1 year
  Time to first AF detected by event recorder transmission will be determined.

SECONDARY OUTCOMES:
number of Emergency room visits/hospitalizations for cardiovascular causes | 1 year
  Subjects will be questioned via telephone interview or clinic visit every 3 months and appropriate hospital recorders retrieved for confirmation of event.
Proportion of patients who develop persistent AF | 1 year
Days in symptomatic AF/Time between successive PAF episodes | 1 year
  The days in which patients report symptomatic AF confirmed by event recorder transmission will be determined and the time interval between successive events will be determined.
AF Severity Scale | 1 year
  Measured via University of Toronto AF Severity Scale at baseline and at end of study or study exit
Adverse effects of assigned therapy | 1 year
  Adverse effects thought to be related to drug therapy will be documented as well as number of patients in whom drug is discontined because of adverse events.
Ventricular rate during AF | 1 year
  Ventricular rate during AF will be measured from the event recorder tracings - from 10 sec of recording
CCS AF Symptom Score | 1 yr
  This will be determined from interview at baseline and each follow-up visit. The CCS AF symptom score is a 5 point score from 0 to 4.
  CCS-SAF Class Definitions
  Class 0 Asymptomatic with respect to AF Class 1 Symptoms attributable to AF have minimal effect on patient's general QOL.
  Class 2 Symptoms attributable to AF have a minor effect on patient's general QOL.
  Class 3 Symptoms attributable to AF have a moderate effect on patient's general QOL.
  Class 4 Symptoms attributable to AF have a severe effect on patient's general QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Gillis, M.D., Principal Investigator — Professor of Medicine
Locations (1):
- University of Calgary, Calgary, Alberta, Canada